CLINICAL TRIAL: NCT06777485
Title: China Liver Cancer Clinical Registry Cohort Database (HEAL)
Status: Recruiting | Type: Observational
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2024KY585
Record Dates: First submitted 2025-01-14; First posted 2025-01-15 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms | interventions — Antineoplastic Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Liver Cancer: Observation of clinical routine treatment in patients with Liver cancer
  Interventions: Procedure: Procedure/Surgery treatment; Drug: Anti-Tumor Drugs

INTERVENTIONS:
Procedure: Procedure/Surgery treatment — Routine surgical operations for patients with hepatocellular carcinoma, such as surgical resection, ablation，TACE，HAIC
Drug: Anti-Tumor Drugs — Use of anti-tumor drugs, e.g., immunologic, targeted, and chemotherapy drugs

SUMMARY:
This study was led by the Department of Hepatobiliary Surgery of the First Affiliated Hospital of the University of Science and Technology of China (USTC), in close cooperation with many participating units across the country, to establish a standardized clinical information database of hepatocellular carcinoma cohorts, which will provide a guarantee for conducting high-quality real-world clinical studies and clinical research.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years, no gender limit
* Patients without surgery are initially diagnosed with hepatocellular carcinoma, intrahepatic cholangiocarcinoma, mixed hepatocellular carcinoma-cholangiocarcinoma, or metastatic hepatocellular carcinoma based on the results of imaging and laboratory tests, or patients with surgery are diagnosed with hepatocellular carcinoma, intrahepatic cholangiocarcinoma, mixed hepatocellular carcinoma-cholangiocarcinoma, or metastatic hepatocellular carcinoma based on the results of pathologic tests
* Signed informed consent, good compliance, willingness to accept follow-up and provide blood and postoperative pathology residual samples

Exclusion Criteria:

* Combination of severe central nervous system disease, respiratory disease, autoimmune disease, chronic renal insufficiency, long-term use of immunosuppressive drugs, combination of severe uncontrolled infections
* Concurrent active cardiovascular disease, cerebrovascular accident within 6 months, myocardial infarction, unstable angina pectoris, or congestive heart failure of class II or greater according to the New York Heart Association criteria, severe arrhythmia requiring medication
* Pregnant or breastfeeding women
* Participation in other therapeutic clinical trials during the course of the patient's illness in which the treatment cannot be specified or information about the treatment cannot be collected

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with hepatocellular carcinoma, intrahepatic cholangiocarcinoma, combined hepatocellular carcinoma-cholangiocarcinoma, or metastatic liver cancer.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2035-01-01 (Estimated); Study Completion 2035-01-01 (Estimated)

PRIMARY OUTCOMES:
OS | 10 years
  Time from enrollment to first recorded occurrence of death from any cause

SECONDARY OUTCOMES:
RFS | 10 years
  Time from enrollment to the first documented occurrence of local, regional, or metastatic liver cancer or death from any cause, whichever occurs first.
Survival time after recurrence | 10 years
  The time from the first documented occurrence of localized, regional, or metastatic liver cancer, whichever occurs first, to death from any cause.

CONTACTS AND LOCATIONS:
Locations (38):
- China (38):
  - Anqing First People's Hospital, Anqing, Anhui
  - Anqing Municipal Hospital, Anqing, Anhui
  - Bengbu First People's Hospital, Bengbu, Anhui
  - The First Affiliated Hospital of Bengbu Medical University, Bengbu, Anhui
  - The Second Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - The People's Hospital of Bozhou, Bozhou, Anhui
  - The People's Hospital of Chizhou, Chizhou, Anhui
  - The First People's Hospital of Chuzhou, Chuzhou, Anhui
  - No.2 People's Hospital of Fuyang City, Fuyang, Anhui
  - Fuyang Cancer Hospital, Fuyang, Anhui
  - Fuyang Fifth People's Hospital, Fuyang, Anhui
  - Fuyang People's Hospital, Fuyang, Anhui
  - Fuyang Sixth People's Hospital, Fuyang, Anhui
  - Funan County People's Hospital, Fuyang, Anhui
  - Taihe County People's Hospital, Fuyang, Anhui
  - Anhui province hospital, Hefei, Anhui
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - Hefei Binhu Hospital, Hefei, Anhui
  - Hefei First People's Hospital, Hefei, Anhui
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - The Second People's Hospital of Hefei, Hefei, Anhui
  - Anhui Second People's Hospital, Hefei, Anhui
  - Huaibei Mining General Hospital, Huaibei, Anhui
  - Huaibei People's Hospital, Huaibei, Anhui
  - Huainan First People's Hospital, Huainan, Anhui
  - Huainan Oriental Hospital, Huainan, Anhui
  - Huainan Sunshine Xinkang Hospital, Huainan, Anhui
  - Huainan Xinhua Hospital, Huainan, Anhui
  - Huangshan City People's Hospital, Huangshan City, Anhui
  - Huangshan Shoukang Hospital, Huangshan City, Anhui
  - Lu'an People's Hospital, Lu'an, Anhui
  - Suzhou Hospital of Anhui Medical University, Suzhou, Anhui
  - Tongling People's Hospital, Tongling, Anhui
  - The Second People's Hospital of Wuhu, Wuhu, Anhui
  - The First Affiliated Hospital of Wannan Medical College, Wuhu, Anhui
  - Xuancheng People's Hospital, Xuancheng, Anhui
  - Henan Provincial People's Hospital, Zhengzhou, Henan

IPD SHARING:
Plan to Share IPD: No